CLINICAL TRIAL: NCT00971451
Title: Quadriceps Function Prior to Anterior Cruciate Ligament Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Joseph M. Hart, Ph.D., Assistant Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13398
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Rupture of Anterior Cruciate Ligament
Keywords: Anterior cruciate ligament; ACL
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Cryotherapy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- knee joint cryotherapy (Experimental): 20 minutes of knee joint cryotherapy - ice bag application
  Interventions: Other: cryotherapy
- TENS (Experimental): continuous TENS for duration of the 1 hour exercise session
  Interventions: Other: TENS
- No intervention (No Intervention): no modality intervention; just exercise

INTERVENTIONS:
Other: cryotherapy — 20 minutes of knee joint cryotherapy - ice bag application
  Arms: knee joint cryotherapy
Other: TENS — continuous use of TENS during the exercise session
  Arms: TENS

SUMMARY:
Patients who are diagnosed with an isolated tear of the anterior cruciate ligament and scheduled for arthroscopic reconstruction using bone-patellar tendon-bone autograft will be recruited to participate.

All subjects will be invited to participate in 2 weeks (2 supervised sessions per week) prior to their surgery. Each session will include supervised therapeutic exercises. Subjects will be randomly assigned to receive continuous transcutaneous electrical nerve stimulation (TENS) during each session or knee joint cryotherapy prior to each exercise session. The investigators will measure quadriceps function before and after this 2-week intervention (both sessions occur prior to reconstruction surgery). This study will also have a true control group that will not receive either exercise of modality intervention. The investigators will collect subjective and objective outcomes data at regularly scheduled post-operative visits.

ELIGIBILITY:
Inclusion Criteria:

1. Complete ACL rupture
2. Age 15-55

Exclusion Criteria:

1. Persons who cannot tolerate knee joint TENS.
2. Persons who have a known allergy to cryotherapy
3. Patients who are pregnant or who plan on getting pregnant during the 12-month follow-up period.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-11; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Quadriceps muscle strength and inhibition using the quadriceps central activation ratio | Day 15

SECONDARY OUTCOMES:
Quadriceps H-reflex testing | Day 15
International Knee Documentation Committee Subjective Knee Joint Evaluation | Day 15
Visual Analog Scale | Day 15
Tegner Activity Rating | Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Hart, Ph.D., Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States